CLINICAL TRIAL: NCT06505109
Title: OPTImizing CArdiac REhabilitation by REfining Sleep and STress
Acronym: OPTICARE-RESST
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Erasmus Medical Center (Other)
Collaborators: Capri Hartrevalidatie (Unknown); Maxima Medical Center (Other); ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, N. (Nienke) ter Hoeve PhD, Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL86677.078.24; 10930012310027 (Other: ZonMw)
Record Dates: First submitted 2024-07-01; First posted 2024-07-17 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Cardiovascular Diseases; Cardiac Rehabilitation
Keywords: Cardiovascular Diseases; Cardiac Rehabilitation; Sleep; Stress
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Intervention Model Description: Patients are randomized to treatment or control.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The intervention group will receive standard CR along with the RESST intervention, consisting of 5-6 on-site group sessions, focused on sleep and stress, integrating principles from Acceptance and Commitment Therapy and Cognitive Behavioral Therapy.
  Interventions: Behavioral: RESST
- Control group (No Intervention): The control group will receive standard CR only. Standard CR programs last around 3-4 months and include two supervised exercise sessions per week. In addition, educational sessions are provided, covering topics such as medical information, cardiovascular risk factors, adopting a heart-healthy lifestyle, and coping with emotions. Depending on the patient's specific needs, counselling sessions on stress management, smoking cessation, and healthy diet are available, and individual counselling can be provided by a social worker, dietician, or psychologist/psychiatrist.

INTERVENTIONS:
Behavioral: RESST — Subjects randomized to the RESST intervention will receive on top of standard rehabilitation a behavioural group intervention focussing on improving sleep and stress. This intervention will consist of 5 till 6 meetings of 90 till 120 minutes in the local rehabilitation centre during a time period of 3 till 4 months.
  Arms: Intervention group

SUMMARY:
The primary objective of this project is to investigate the effectiveness and costs of integrating a behavioural program targeting sleep and stress (the RESST intervention) into cardiac rehabilitation (CR). In addition, the investigators will also study whether parameters regarding diversity (e.g., sex, ethnicity, socioeconomic position) are associated with intervention effectiveness. Furthermore, the investigators aim to explore the (bidirectional) relation between sleep and stress on the one hand, and other lifestyle components and health outcomes on the other hand.

DETAILED DESCRIPTION:
CR focuses on the secondary prevention of cardiovascular disease (CVD) by promoting a healthy lifestyle and is a valuable approach to improve quality of life, mortality and hospital readmissions. However, optimization of CR is necessary. Current CR programs pay insufficient attention to sleep and stress problems, despite more than 50% of CVD patients experiencing sleep problems and high stress levels. Both sleep and stress are associated with adverse cardiovascular health and a decreased quality of life. The hypothesis for this study is that adding a behavioural intervention will improve sleep and perceived stress (primary outcomes), along with positive outcomes on biomarkers of chronic stress, QoL, cardiometabolic risk factors, physical fitness, lifestyle components, and psychosocial well-being.

The project involves a multicenter randomized controlled trial. The intervention group (100 patients) will receive standard CR along with the RESST intervention, consisting of 5-6 on-site group sessions integrating principles from Acceptance and Commitment Therapy and Cognitive Behavioral Therapy and focused on improving sleep and stress. The control group (100 patients) will receive standard multidisciplinary CR only.

The primary outcomes of the study include both objective and subjective measures of sleep, as well as perceived stress. Secondary outcomes encompass quality of life, chronic stress biomarkers, cardiometabolic risk factors, physical fitness, lifestyle components and psychosocial wellbeing. These outcomes will be assessed before and after the intervention, as well as at a 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age at or above 18 years
* Proficient in the Dutch language
* Experiencing sleep and/or stress problems as indicated by a high score on the Pittsburgh Sleep Quality Index (PSQI score >5) or Perceived Stress Scale-10 (PSS-10 score >13)
* Signed informed consent

Exclusion Criteria:

* Severe psychiatric, cognitive or physical comorbidity that would impede CR participation
* Active treatment for sleep disorders, stress, or other forms of (behavioural) therapy at the start of the study or expected to start within the first 6 months of the study, that could interfere with the RESST intervention. Note: Participants with previously diagnosed sleep disorders are eligible if they still experience sleep or stress problems, unless they fall under the above criteria. Participants who received a prior treatment that is still ongoing but has resulted in a stable sleep and stress condition in the 3 months before the cardiovascular event (e.g., Continuous Positive Airway Pressure (CPAP)) are eligible.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-08-28 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Objectively assessed sleep duration | At baseline, after 3 months, and after 6 months.
  This will be measured with a GENEACTIV accelerometer for 7 days and nights continuously.
Objectively assessed sleep-onset latency | At baseline, after 3 months, and after 6 months.
  This will be measured with a GENEACTIV accelerometer for 7 days and nights continuously.
Objectively assessed wake after sleep onset | At baseline, after 3 months, and after 6 months.
  This will be measured with a GENEACTIV accelerometer for 7 days and nights continuously.
Objectively assessed sleep efficiency | At baseline, after 3 months, and after 6 months.
  This will be measured with a GENEACTIV accelerometer for 7 days and nights continuously.
Self-reported sleep quality | At baseline, after 3 months, and after 6 months.
  This will be measured with the Pittsburgh Sleep Quality Index (PSQI) questionnaire. Score between 0-21, higher score indicates worse sleep quality.
Perceived stress level | At baseline, after 3 months, and after 6 months.
  This will be measured with the Perceived Stress Scale-10 (PSS-10) questionnaire. Score between 0-40, higher score indicates higher perceived stress.

SECONDARY OUTCOMES:
Cortisol level | At baseline, after 3 months, and after 6 months.
  This will be measured by taking a hair sample. The amount of cortisol in the hair will be determined in a lab.
Cortisone level | At baseline, after 3 months, and after 6 months.
  This will be measured by taking a hair sample. The amount of cortisone in the hair will be determined in a lab.
Weight | At baseline, after 3 months, and after 6 months.
  Weight will be measured with a digital scale in kilograms.
Height | At baseline.
  Height will be measured with a stadiometer in centimeters.
Body Mass Index (BMI) | At baseline, after 3 months, and after 6 months.
  Weight and height will be combined to report BMI in kg/m^2.
Blood pressure | At baseline, after 3 months, and after 6 months.
  Blood pressure will be measured with a blood pressure monitor.
Smoking behaviour | At baseline, after 3 months, and after 6 months.
  This will be measured with a carbon monoxide breath tester.
Smoking behaviour | At baseline, after 3 months, and after 6 months.
  This will be measured with a self-designed questionnaire. The outcome of this questionnaire indicates whether a person smokes/has smoked in the past/does not smoke, what sort of tobacco is being smoked and how much the participant smokes.
Muscle strength | At baseline, after 3 months, and after 6 months.
  Handgrip strength will be measured with a hand dynamometer.
Physical activity | At baseline, after 3 months, and after 6 months.
  This will be measured with a GENEACTIV accelerometer for 7 days and nights continuously.
Sedentary behaviour | At baseline, after 3 months, and after 6 months.
  This will be measured with a GENEACTIV accelerometer for 7 days and nights continuously.
Alcohol use | At baseline, after 3 months, and after 6 months.
  This will be measured with the five-shot questionnaire. Score between 0-7, higher score indicates higher chance of alcohol overuse, misuse, and dependency.
Health related quality of life | At baseline, after 3 months, and after 6 months.
  This will be measured with the MacNew questionnaire. Score between 1-7, higher score indicates higher health related quality of life.
Health related quality of life | At baseline, after 3 months, and after 6 months.
  This will be measured with the EuroQol 5D/EQ5D questionnaire. Score between -0.446 - 1, higher score indicates a better health state. One subscale has a score between 0-100, higher score indicates better perceived health.
Fatigue | At baseline, after 3 months, and after 6 months.
  This will be measured with the Fatigue Severity Scale (FSS) questionnaire. Score between 9-63, higher score indicates a greater fatigue severity.
Daytime sleepiness | At baseline, after 3 months, and after 6 months.
  This will be measured with the Epworth Sleepiness Scale (ESS) questionnaire. Score between 0-24, higher score indicates a higher level of daytime sleepiness.
Anxiety and depression | At baseline, after 3 months, and after 6 months.
  This will be measured with the Hospital Anxiety and Depression Scale (HADS) questionnaire. Score between 0-21 per subscale, higher score indicates severe symptoms of anxiety and depression.
Participation in society | At baseline, after 3 months, and after 6 months.
  This will be measured with the USER-Participatie (USER-P) questionnare. Score between 0-100, higher score indicates higher participation in society.
Estimated Cardiorespiratory fitness | At baseline, after 3 months, and after 6 months.
  This will be measured with the FitMáx©-Questionnaire. The outcome of this questionnaire is the estimated maximum oxygen uptake expressed in mL/kg/min. Higher score indicates better cardiorespiratory fitness.
Presence of restless leg syndrome | At baseline.
  This will be measured with the RLS rating scale questionnaire. Score between 0-28, higher score indicates more severe symptoms of restless leg syndrome.
Presence of insomnia | At baseline.
  This will be measured with the Insomnia Severity Index (ISI) questionnaire. Score between 0-28, higher score indicates more severe insomnia complaints.
The risk of the presence of obstructive sleep apnoea | At baseline.
  This will be measured with the STOP-bang questionnaire. Score between 0-8, higher score indicates higher risk of obstructive sleep apnoea.
Costs incurred by the patients | After 3 months and after 6 months.
  This will be measured with the IMTA Medical Consumption Questionnaire (IMCQ) which aims to determine costs within the health care system.
Productivity costs | After 3 months and after 6 months.
  This will be measured with the IMTA Productivity Costs Questionnaire (IPCQ) which aims to determine the cost of productivity losses.
Perceived sleep | At baseline, after 3 months, and after 6 months.
  This will be measured with the Sleep Consensus Diary for 7 days. The Sleep Consensus Diary consists of questions about the experience of sleep, what time the participant went to sleep, and how often the participant woke up.
Diet | At baseline, after 3 months, and after 6 months.
  This will be measured with an electronic diary. Intake of caffeine and alcohol and timing of the main meal will be measured.
Momentary fatigue | At baseline, after 3 months, and after 6 months.
  This will be measured with an electronic diary.
Momentary stress | At baseline, after 3 months, and after 6 months.
  This will be measured with an electronic diary.
Adherence to the CR treatment and RESST intervention | After 3 months.
  This will be measured by recording the number of rehabilitation components attended, such as courses on nutrition or personal counseling.
Treatment Satisfaction | After 3 months.
  This will be measured with a self-designed questionnaire and consists of questions about the applicability, clarity and logistics of the intervention.
Sex | At baseline.
  Female / male / other
Age | At baseline.
  Age in years.
Cardiac diagnosis | At baseline.
  Cardiac diagnosis as defined by ICD-10 that has resulted in referral to cardiac rehabilitation.
Educational level | At baseline.
  Single-item question (high, middle, or low educated).
Relational status | At baseline.
  Single-item question.
Cardiac risk factors | At baseline.
  Presence of cardiac risk factors (family history, diabetes mellitus, hypertension, dyslipidemia, smoking prior to event).
Cardiac history | At baseline.
  History of cardiovascular events and diseases.
Medication usage | At baseline, after 3 months, and after 6 months.
  Number of participants using a certain type of prescribed and/or over-the-counter medication.
Comorbidity | At baseline.
  Presence of other diseases.
Socioeconomic status | At baseline.
  Socioeconomic status indicated by postal code.
Origin | At baseline.
  Determined by birth country and parents' birth country.
Employment | At baseline.
  Determined by employment status, and type of job.
Drug use | At baseline.
  Drug use (yes/no) and drug classification.
Current/previous sleep disorder treatment | At baseline.
  Description of current and previous treatment for sleeping disorders.

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Máxima Medisch Centrum, Eindhoven, North Brabant
  - Capri Hartrevalidatie, Rotterdam, South Holland
  - Capri Hartrevalidatie, The Hague, South Holland

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: After termination of the study.
Access Criteria: The processed data will be made available in a repository. The Principal investigator can be contacted to request access to the data. Access to the data is evaluated by the OPTICARE RESST Consortium. If allowed based on the consortium agreement and the informed consent and when the intended methodology seems suitable data can be shared after signing of a DTA. Data will be further pseudonymized before sharing.